CLINICAL TRIAL: NCT01851629
Title: Adaptive Walking Responses Critical for Effective Community Ambulation Post-Incomplete Spinal Cord Injury
Brief Title: Walking Adaptability Post-Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Malcom Randall VA Medical Center (U.S. Federal Agency); James A. Haley Veterans Administration Hospital (U.S. Federal Agency); Brooks Rehabilitation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 01-2013; W81XWH-11-1-0454 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2013-04-24; First posted 2013-05-10 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Incomplete Spinal Cord Injury; Brown Sequard Syndrome
Keywords: Locomotor training; Walking recovery; Neuroplasticity
MeSH Terms: conditions — Brown-Sequard Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ADAPT Locomotor Training (Experimental): Individuals receive 15 sessions of ADAPT-locomotor training for 3 weeks. During ADAPT-locomotor training, stepping in response to obstacles and walking challenges are practiced on a treadmill and overground.
  Interventions: Behavioral: Locomotor Training
- Basic Locomotor Training (Active Comparator): Individuals will receive 15sessions of the traditional form of basic locomotor training for 3 weeks. Repetitive stepping patterns are practiced on the treadmill and overground.
  Interventions: Behavioral: Locomotor Training
- Cross-Sectional Testing (Other): Individuals with and without spinal cord injury will be evaluated to develop protocols within our laboratory to assess reflexes (spinal tract integrity), walking ability, and whether mirror images during walking enhance or disrupt motor responses during walking.
  Interventions: Other: Cross-Sectional Testing (No Intervention)

INTERVENTIONS:
Behavioral: Locomotor Training — Individuals are provided manual assistance for intense, task-specific stepping practice on a treadmill and overground.
  Arms: ADAPT Locomotor Training; Basic Locomotor Training
Other: Cross-Sectional Testing (No Intervention) — Individuals with and without spinal cord injury will be evaluated to develop protocols within our laboratory to assess reflexes (spinal tract integrity), walking ability, and whether mirror images during walking enhance or disrupt motor responses during walking.
  Arms: Cross-Sectional Testing

SUMMARY:
The purpose of this study is: (1) to establish assessment techniques (in our laboratory) to identify the functional integrity of long spinal tracts associated with adaptive walking recovery post-spinal cord injury and (2) to preliminary investigate locomotor outcomes associated with an adaptive locomotor training approach post-spinal cord injury.

DETAILED DESCRIPTION:
Eligible individuals without spinal cord injury that are enrolled in the study will participate for 1-2 days. These individuals may undergo a variety of non-invasive neurophysiological tests which evaluate spinal reflexes and integrity of specific spinal pathways. In addition, their movement may be assessed during walking on a treadmill and overground in a variety of different conditions (e.g. with mirrors, without mirrors, with obstacles, without obstacles).

Eligible individuals with spinal cord injury that are enrolled in the study will undergo the same testing as described above for the healthy controls. In addition, a small subset of these individuals may receive locomotor training (3 weeks of basic locomotor training followed by 3 weeks of adaptive locomotor training, separated by a 3 week washout period). For the individuals receiving locomotor training, they will be tested before and after each 3 week training session.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* no neurologic injury (for individuals without SCI)
* >12 mos post-incomplete SCI (iSCI), discharged from in- and out-patient rehabilitation, with diagnosis of first time motor iSCI (AIS C or D with upper motor neuron lesions at cervical or thoracic levels) (for individuals with SCI)
* medically stable condition with no changes in anti-spasticity meds
* ability to walk in the home and/or ambulate in the community using a single cane or crutch, bilateral canes or crutches, or no device
* walking speeds > 0.3 m/sec, with deficit performance on the Dynamic Gait Index
* medically approved for participation

Exclusion Criteria:

* current participation in another rehabilitation program/research protocol
* history of congenital SCI or other degenerative spinal disorders
* inappropriate or unsafe fit of the harness and/or joint contractures or severe spasticity that would prohibit the safe provision of training
* receipt of a therapeutic intervention or medication within the last 6 mos that would alter the nervous system's ability to respond to treatment (e.g. Botox injections)
* unable to safely receive transcranial magnetic stimulation due to positive history which prohibits its use

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-06; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Changes in joint movement (Kinematics) | At approximately 0 weeks (pre-LT#1), 3 weeks (post-LT#1), 6 weeks (pre-LT#2) and 9 weeks (post-LT#2). Times may vary slightly if training sessions are missed (i.e. due to illness).
  During walking on the treadmill and overground, movement of lower extremity joints (hip, knee, and ankle) will be quantified using reflective markers and a 3D motion analysis system.

SECONDARY OUTCOMES:
Changes in falls risks during adaptive walking challenges | At approximately 0 weeks (pre-LT#1), 3 weeks (post-LT#1), 6 weeks (pre-LT#2) and 9 weeks (post-LT#2). Times may vary slightly if training sessions are missed (i.e. due to illness).
  Individuals will be tested on a special treadmill that perturbs walking and makes indirect measurements related to falls risks
Changes in functional integrity of spinal pathways | At approximately 0 weeks (pre-LT#1), 3 weeks (post-LT#1), 6 weeks (pre-LT#2) and 9 weeks (post-LT#2). Times may vary slightly if training sessions are missed (i.e. due to illness).
  Non-invasive protocols will be used to test a variety of reflexes that provide indirect measures related to the integrity of specific spinal pathways.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole J Tester, PhD, Principal Investigator — University of Florida; Emily J. Fox, PhD, DPT, NCS, Principal Investigator — University of Florida; Carolynn Patten, PhD, PT, Principal Investigator — University of Florida
Locations (4):
- United States (4):
  - University of Florida, Gainesville, Florida
  - Brain Rehabilitation Research Center, Malcom Randall VAMC, Gainesville, Florida
  - Brooks Rehabilitation, Jacksonville, Florida
  - James A. Haley VA Medical Center, Tampa, Florida